CLINICAL TRIAL: NCT01415908
Title: A Prospective, Multi-center, Pivotal Trial for INFUSE® Bone Graft With CAPSTONE® Spinal System and Posterior Supplemental Fixation to Treat 1- or 2-level Advanced Degenerative Disease of the Lumbosacral Spine For a TLIF Approach
Brief Title: INFUSE®Bone Graft in Transforaminal Lumbar Interbody Fusion for Degenerative Disease of Lumbosacral Spine
Acronym: TLIF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to study design challenges including DMC enrollment suspension as required by the protocol stopping rules and recommended changes to the surgical technique
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medtronic P05-06
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Lumbar Spine Degeneration
Keywords: advanced degenerative disease of the lumbosacral spine; lumbosacral spine; radiculopathy; degenerative instability; spondylolisthesis; retrolisthesis; lateral listhesis; spinal stenosis; disc herniation; INFUSE Bone Graft; CD HORIZON Spinal System; CAPSTONE Spinal System
MeSH Terms: conditions — Radiculopathy; Spondylolisthesis; Spinal Stenosis; Intervertebral Disc Displacement | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Iliac Crest Bone Graft
- Investigational Group (Experimental)
  Interventions: Device: INFUSE Bone Graft

INTERVENTIONS:
Device: INFUSE Bone Graft — Subjects enrolled in the investigational treatment group will receive surgical treatment with INFUSE® Bone Graft, the CAPSTONE® Spinal System, and posterior supplemental fixation (in this study the CD HORIZON® Spinal System). The investigational treatment will be implanted using a TLIF surgical approach.
  Other Names: rhBMP-2/ACS; Dibotermin alfa
  Arms: Investigational Group
Other: Iliac Crest Bone Graft — Subjects enrolled in the control group will receive the same surgical treatment as the investigational group, including the CAPSTONE® Spinal System and posterior supplemental fixation system (CD HORIZON® Spinal System), except for the use of autogenous bone graft (from the iliac crest) instead of INFUSE® Bone Graft. A TLIF surgical approach will also be used for implanting the control treatment.
  Other Names: Autograft
  Arms: Control Group

SUMMARY:
This investigation will provide safety and effectiveness information on the use of INFUSE® Bone Graft with the CAPSTONE® Spinal System and CD HORIZON® Spinal System with a Transforaminal Lumbar Interbody Fusion (TLIF) surgical approach at one or two adjacent levels from L2-S1 to treat subjects with advanced degenerative disease of the lumbosacral spine.

DETAILED DESCRIPTION:
The study is a prospective, multi-national study that compares INFUSE® Bone Graft (investigational group) to autogenous bone graft (control group). Control group subjects will receive the same surgical treatment except for the use of autogenous bone graft (from the iliac crest) instead of INFUSE® Bone Graft. All sites will follow a common Clinical Investigational Plan (CIP) that consists of the protocol and accompanying case report forms, risk analysis, investigator's agreement, subject informed consent, institutional review board (IRB) certification, labeling, and monitoring information.

ELIGIBILITY:
Inclusion Criteria:

* Has advanced degenerative disease of the lumbosacral spine (L2 to S1) that results in radiculopathy secondary to nerve root compression, manifested by, History of radiating leg or buttock pain, paresthesias, numbness or weakness, or History of neurogenic claudication.
* Has a history of low back pain
* Has radiographic evidence of advanced degenerative lumbosacral disease, such as decreased disc height; herniated nucleus pulposus; hypertrophy or thickening of the ligamentum flavum, annulus fibrosis, or facet joint capsule; hypertrophied facet joints, facet joint space narrowing, or facet periarticular osteophyte formation; trefoil canal shape; or lateral(subarticular) stenosis; or vertebral endplate osteophyte formation; and at least one of the following:

Sagittal plane translation (slippage) of the superior (cranial) vertebral body anterior or posterior to the inferior (caudal) vertebral body greater than 3mm, or Coronal plane translation (slippage) of the superior (cranial) vertebral body lateral to the inferior (caudal) vertebral body greater than 3mm, or Narrowing (stenosis) of the lumbar spinal canal and/or intervertebral foramen

* Has single-level or adjacent two-level involvement from L2 to S1.
* Has preoperative Oswestry score ≥30.
* Has preoperative back pain score of ≥ 6 based on the Preoperative Back and Leg Pain Questionnaire (pain intensity + pain frequency).
* Has preoperative leg pain score of ≥ 6 based on the Preoperative Back and Leg Pain Questionnaire (pain intensity + pain frequency).
* Is at least 18 years of age and skeletally mature at the time of surgery.
* Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of six months.
* Is willing and able to comply with the study plan and able to understand and sign the Subject Informed Consent Form.

Exclusion Criteria:

* Requires spinal fusion at more than two lumbar levels or at two non-adjacent levels.
* Has had a prior lumbar surgical fusion procedure at the involved or adjacent spinal levels.
* Has significant lumbar instability, defined as sagittal or coronal plane listhesis greater than Grade 2 spondylolisthesis utilizing Meyerding's Classification (Meyerding, HW, 1932).
* Has scoliosis greater than 30 degrees.
* Has had a previous diagnosis of osteoporosis, osteopenia, or osteomalacia.
* In addition, if the subject has any of the following risk factors, a DEXA scan should be performed to determine eligibility:

History of a non-traumatic hip or spine fracture. Female who is postmenopausal. Female over the age of 65. Male over the age of 70. If the DEXA T-score is -2.5 or lower, OR a T-score of -1.5 or lower WITH a history of a vertebral compression fracture, the subject is excluded.

* Is morbidly obese, as defined as a Body Mass Index (BMI) > 40.
* Has an active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
* Has an overt or active bacterial infection, either local or systemic.
* Has undergone systemic administration of any type of corticosteroid, anti-neoplastic, immunostimulating, or immunosuppressive agents within 30 days prior to implantation of the assigned treatment.
* Has a history of clinically significant cardiac or hematologic disease.
* Has a history of autoimmune disease known to affect bone metabolism or the spine. Examples include spondyloarthropathies (e.g., ankylosing spondylitis, Crohn's disease, and ulcerative colitis), juvenile arthritis, rheumatoid arthritis, Grave's disease, and Hashimoto's thyroiditis.
* Has a medical disease or condition that would preclude accurate clinical evaluation of the safety and effectiveness of the treatments in this study, such as motor weakness, sensory loss, or painful conditions that inhibit normal ambulation or other activities of daily living.
* Has a history of any endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).
* Has chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease.
* Has a history of exposure to injectable collagen.
* Has received any previous exposure to any/all BMPs of either human or animal extraction.
* Has a history of hypersensitivity to collagen or protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins).
* Has a history of any allergy resulting in anaphylaxis.
* Has a history of allergy to bovine products.
* Has a documented allergy or intolerance to titanium, titanium alloy, tantalum, tantalum alloy, or polyetheretherketone (PEEK).
* Has any condition in which MRI scans are contraindicated (e.g., cardiac pacemaker, brain aneurysm clips).
* Has any condition in which a gadolinium-contrast MRI is contraindicated (e.g., sickle cell anemia, renal failure).
* Is mentally incompetent. If questionable, obtain psychiatric consult.
* Has a 'Waddell Signs of Inorganic Behavior' score of 3 or greater.
* Is a prisoner.
* Is a tobacco user who does not agree to suspend tobacco use prior to surgery.
* Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
* Has received treatment with an investigational therapy (drug, device and/or biologic) within 28 days prior to implantation surgery or such treatment is planned during the 24-month period following the study surgery.
* Is pregnant or nursing. Female of child-bearing potential must agree not to become pregnant for one year following surgery.
* Is a Worker's Compensation case or is involved in spinal litigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sonoran Spine Center, Mesa, Arizona
  - USC Department of Neurological Surgery, Los Angeles, California
  - Andrews Institute, Gulf Breeze, Florida
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - UPMC Presbyterian, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Group: Investigational subjects received INFUSE® bone graft, with the CAPSTONE® Spinal System and posterior supplemental fixation (CD HORIZON® Spinal System) using TLIF surgical approach.
- Control Group: Control subjects received autogenous bone graft from iliac crest, with CAPSTONE® Spinal System and posterior supplemental fixation system (CD HORIZON® Spinal System) using TLIF surgical approach.
Period: Overall Study
Arm/Group | Investigational Group | Control Group
Started | 11 | 4
Completed | 10 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group | Control Group | Total
Number analyzed (Participants) | 11 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.88) | 56.2 (12.26) | 52.0 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9 | 4 | 13
  Black | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Hispanic | 0 | 0 | 0
  Other | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Inches] | 67.6 (3.35) | 68.5 (3.87) | 67.9 (3.38)
Weight [Mean (Standard Deviation); unit: lbs] | 179.7 (37.25) | 183.5 (38.10) | 180.7 (36.13)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Success
Description: Rate of overall success is reported as percent of subjects who met all of the following criteria:
  1. fusion at all treated levels (e.g., one level for a one level fusion and two levels for a two level fusion);
  2. pain/disability (Oswestry Disability Index) success;
  3. neurological status success;
  4. no serious adverse event classified as "implant associated" or "implant/surgical procedure associated";
  5. no additional surgical procedure classified as a "failure."
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants | 70.0 | 50.0

2. Secondary Outcome: Rate of Fusion Success
Description: Rate of fusion success is reported as percent of subjects having fusion success. The fusion success was defined radiologically as:
  1. evidence of bridging bone;
  2. no evidence of motion;
  3. no evidence of radiolucency at greater than 50% of the superior or inferior PEEK spacer-vertebra interface.
Time Frame: 24 months
Population: Eight investigational and 3 control subjects were evaluated for fusion success at 24 months.
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 8 | 3
percentage of participants | 100.0 | 100.0

3. Secondary Outcome: Success Rate of Oswestry Disability Index
Description: ODI Questionnaire was used to assess patient back function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability). Success rate of Oswestry Disability Index (ODI) is reported as percent of subjects whose ODI score met: pre-operative score - post-operative score ≥ 15.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants | 90.0 | 75.0

4. Secondary Outcome: Success Rate of Neurological Status
Description: Neurological status was assessed in six sections: motor, sensory, reflexes, straight leg raising, bowel function, and bladder function. Each of the sections had a number of elements. Success rate of neurological status is reported as percent of subjects whose neurological status was maintained or improved in three key neurological assessments-motor, sensory, and deep tendon reflexes.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants | 80.0 | 50.0

5. Secondary Outcome: Success Rate of Back Pain
Description: Numerical rating scales were used to evaluate back pain intensity and frequency. Subjects rated their back pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, subjects recorded their back pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total back pain score were the sum of pain intensity and frequency scores. Success rate of back pain is reported as percent of subjects whose back pain improvement met: pre-operative score - post-operative score > 0.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants | 100.0 | 100.0

6. Secondary Outcome: Success Rate of Leg Pain
Description: Numerical rating scales were used to evaluate leg pain intensity and frequency. Subjects rated their leg pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, subjects recorded their leg pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." The total leg pain score were the sum of pain intensity and frequency scores. Success rate of leg pain is reported as percent of subjects whose leg pain improvement met: pre-operative score - post-operative score > 0.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants | 90.0 | 100.0

7. Secondary Outcome: Success Rate of General Health Status
Description: The Medical Outcomes Study 36-Item Short Form (SF-36) health survey was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The scores for PCS and MCS are between 0 and 100, with higher scores denoting better quality of life. To be classified as a success, the following criteria must be met for SF-36 PCS and MCS, respectively: post-operative score - pre-operative score >= 0. The results are reported as percent of subjects who have SF-36 PCS success, SF-36 MCS success, and overall SF-36 success.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 10 | 4
percentage of participants
  Overall SF-36 success | 70.0 | 75.0
  Success of SF-36 PCS | 80.0 | 100.0
  Success of SF-36 MCS | 80.0 | 75.0

8. Secondary Outcome: Percent of Subjects Who Had Additional Surgical Procedures/Interventions
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 11 | 4
percentage of participants | 18.2 | 50.0

9. Secondary Outcome: Operative Time
Time Frame: Operative time was recorded from skin incision to wound closure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 11 | 4
minutes | 200.0 (114.24) | 281.5 (38.17)

10. Secondary Outcome: Blood Loss
Time Frame: During the operation, an average of 200 minutes for investigational group and 281.5 minutes for control group
Measure: Mean (Standard Deviation); unit: mls
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 11 | 4
mls | 322.7 (267.73) | 200.0 (191.49)

11. Secondary Outcome: Hospital Stay
Time Frame: During the time of hospital stay
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Investigational Group | Control Group
Number analyzed (Participants) | 11 | 4
days | 4.2 (1.17) | 4.5 (1.00)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Investigational Group | Control Group
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/4
Other Adverse Events (participants affected / at risk) | 9/11 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=11) | Control Group (N=4)
post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group (N=11) | Control Group (N=4)
haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
oedema peripheral (General disorders) | 1 (1) | 0 (0)
pyrexia (General disorders) | 2 (3) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (2) | 0 (0)
dural tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
vitamin D decreased (Investigations) | 1 (1) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (2)
hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 1 (2) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hot flush (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A total of 534 ± 10 subjects were planned for enrollment. However, this study was terminated early with only 15 enrolled patients, leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less